CLINICAL TRIAL: NCT04364646
Title: Personalized Integrated Chronotherapy for Perinatal Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: Northwell Health (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Katherine M. Sharkey, Principal Investigator, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-0913
Record Dates: First submitted 2020-04-06; First posted 2020-04-28 (Actual); Results first posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Depression; Postpartum Depression; Prenatal Disorder; Circadian Dysregulation; Pregnancy Related; Sleep Disturbance
MeSH Terms: conditions — Depression; Depression, Postpartum; Chronobiology Disorders; Parasomnias | interventions — Chronotherapy; Ultraviolet Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: outcome assessments are made by a blinded investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Women in the usual care group receive medications and/or talk therapy. Sleep and light levels are monitored at home with wrist actigraphy during 3rd trimester of pregnancy (weeks 28-40) and weeks 2-6 and18 after the baby is born (postpartum weeks 2-6 and 18).
  Interventions: Behavioral: Personalized Integrated Chronotherapy
- Personalize Integrated Chronotherapy (Experimental): Women in the integrated chronotherapy group receive usual care (medications and/or talk therapy, as above) and also receive a bright light box to sit with every morning for up to 60 minutes as prescribed by the study doctor.
  Interventions: Behavioral: Personalized Integrated Chronotherapy

INTERVENTIONS:
Behavioral: Personalized Integrated Chronotherapy — Based on their baseline sleep-wake schedule and real-life constraints (work and other responsibilities), an initial sleep schedule is set that allows 7.5 hours of sleep and provides time for participants to sit in front of the morning bright light.
  Other Names: Chronotherapy; Triple Chronotherapy; Bright Light Therapy

SUMMARY:
Perinatal depression and anxiety are common, serious, and frequently overlapping disorders that increase morbidity and mortality in new mothers (including suicide) and result in poor infant/child outcomes. Current therapies often fail to produce recovery or are poorly tolerated, and many pregnant women seek non-pharmacologic therapy or forgo treatment when non-pharmacologic options are not available. Expectant and new mothers who experience circadian rhythm dysregulation are at increased risk for perinatal depression. This Confirmatory Efficacy Clinical Trial of Non-Pharmacological Interventions for Mental Disorders R01 seeks to test whether a Personalized Integrated Chronotherapy (PIC) intervention can improve treatment outcomes for pregnant patients seeking outpatient treatment for depression, with or without anxiety. PIC is a multicomponent treatment consisting of bright light therapy, sleep phase advance, and sleep stabilization/restriction that targets the Research Domain Criteria (RDoC) constructs of circadian rhythms and sleep-wake behavior. To increase sample size and diversity and accelerate recruitment, this study will be performed at 4 sites that differ in clinical structure and that have piloted the PIC intervention. The study will enroll expectant mothers diagnosed with major depressive disorder during 3rd trimester of pregnancy. Participants will be randomized to either: (a) usual care (UC, n = 110) or (b) PIC+UC (n = 110). PIC+UC will have pregnancy and postpartum components and will be administered via a personalized approach tailored to optimize the intervention based on each patient's individual circadian and sleep timing. After a baseline assessment, PIC will be prescribed during 5 dedicated clinical visits: three during 3rd trimester of pregnancy and 2 in the postpartum period. UC will consist of medication and/or psychotherapy. UC will be quantified in both groups to evaluate differences between the PIC+UC and UC groups. Mood will be measured in both groups by blinded clinician interview and patient self-report. The safety profile of the PIC intervention will be assessed by evaluation of side effects/adverse events. Importantly, the study will also examine the target mechanisms by which PIC is hypothesized to work and test the mediation effects of the circadian targets on improvement in mood symptoms. Participants will wear wrist actigraphy/light monitors continuously during weeks 28-40 of pregnancy and postpartum weeks 2-6 to assess light exposure and to estimate sleep timing and duration. Circadian phase (measured with salivary dim light melatonin onset) will be measured at baseline during pregnancy (~30 weeks' gestation), at 36 weeks' gestation, and at postpartum week 6. Exploratory aims will examine associations between infant sleep behavior and maternal circadian rhythms and factors relevant to future dissemination of PIC. If this intervention is effective, perinatal PIC could change clinical practice and have major public health impact due to the high prevalence of perinatal depression and anxiety, the negative effects of mood disorders on mothers and their children, and the need to provide effective, novel, non-pharmacologic therapies for women with perinatal mood disorders.

DETAILED DESCRIPTION:
The purpose of this research study is to collect data on whether adding light therapy and a prescribed sleep schedule to usual treatment for depression can reduce depression and anxiety symptoms during pregnancy and the postpartum. The study is enrolling pregnant woman between the ages of 18 and 40 who have been diagnosed with depression and (possibly) anxiety.

This study takes place from the 3rd trimester of pregnancy to 18 weeks postpartum. Women who take part in this study will be randomly assigned ("randomized") into one of the study treatment groups (1) the "usual care" group (UC); or (2) the group that receives bright light therapy and a prescribed sleep schedule, also called the "Personalized Integrated Chronotherapy" group (PIC). The usual care group will receive medications and/or talk therapy as decided by the woman and her doctor. Women in the integrated chronotherapy group will receive usual care (as above) and will also receive a bright light box to sit with every morning for up to 60 minutes as prescribed by the study doctor. Light will be delivered with a portable, broad-spectrum light box. Both groups will have their sleep and light levels monitored during 3rd trimester of pregnancy (weeks 28-40) and weeks 2-6 and 18 after the baby is born (postpartum weeks 2-6 and 18) Sleep monitoring takes place in the home using a small wrist activity monitor called an "actigraph." Participants will also be asked to provide three saliva sample sets over the course of the study to measure melatonin levels.

In addition to the "Personalized Integrated Chronotherapy" study treatment that will supplement the clinical care as described above, participants will be asked to come in for research study visits.

ELIGIBILITY:
Inclusion Criteria:

- pregnant women, ages 18-45 years with a HAMD score >=14 and a current DSM-5 diagnosis of major depressive disorder as determined with the Current Major Depression Module of the Structured Clinical Interview for DSM disorders (SCID-I/P)

Exclusion Criteria:

* active psychosis or suicidality contraindicating outpatient treatment as determined by the clinical judgement of the research team and as measured with the B/C module of the SCID-I/P and the Columbia-Suicide Severity Rating Scale
* bipolar disorder (because sleep restriction can increase risk of conversion to mania)
* seizure disorder (because sleep restriction can increase seizure risk)
* self report of frequent migraines/headaches precipitated by bright light or sleep deprivation
* preexisting eye/skin disorders contraindicating light therapy
* use of photosensitizing medications
* primary Axis I diagnosis other than MDD (e.g., anorexia nervosa, ADHD)
* high risk pregnancy (e.g., conditions requiring mandatory bed rest or complex medical regimens that will interfere with study participation or conditions where poor infant outcomes are anticipated)
* starting antidepressants in the 4 weeks prior to enrollment
* current employment as night shift worker
* Alcohol Use Disorders Identification Test (AUDIT) score > 8 and/or Drug Abuse Screening Test (DAST) > 1 indicating current alcohol or drug use disorders
* women whose infants will not be living in the home or who will have a nighttime caregiver
* Pittsburgh Sleep Quality Inventory (PSQI)190 < 5 (i.e., those who report no sleep complaints during 3rd trimester of pregnancy and for whom an intervention targeting sleep might not be indicated).
* women who do not speak and read English because PIC research instruments are only available in English at this time. If this RCT shows effectiveness, future work will examine effectiveness in women who speak and read languages other than English.
* Women who experience fetal loss or stillbirth, as well as mothers whose infants are born before 36 weeks' gestation or have NICU stays > 5 days, will be discontinued from the study but will continue to receive UC.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — people who can become pregnant are eligible, i.e., female sex; any gender identity can be enrolled but must be pregnant
Enrollment: 120 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2025-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristina M Deligiannidis, MD, Principal Investigator — Northwell Health; Samantha Meltzer-Brody, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (3):
- United States (3):
  - Feinstein Institute For Medical Research, Glen Oaks, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Rhode Island Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
Per NIMH guidelines
Supporting Information: Study Protocol, CSR
Time Frame: when study is concluded and data are prepared
Access Criteria: with approval from PI and regulatory bodies

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | Personalize Integrated Chronotherapy
Started | 63 | 57
Completed | 51 | 38
Not Completed | 12 | 19
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 7 | 14
Not completed — Protocol Violation | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Personalize Integrated Chronotherapy | Total
Number analyzed (Participants) | 63 | 57 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 63 | 57 | 120
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (4.4) | 31.8 (4.8) | 32.4 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 57 | 120
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 10 | 18
  Not Hispanic or Latino | 55 | 46 | 101
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 9 | 9 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 6 | 18
  White | 35 | 37 | 72
  More than one race | 4 | 5 | 9
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 63 | 57 | 120
Hamilton Depression Rating Scale Score [Mean (Standard Deviation); unit: units on a scale] — (The Hamilton Depression Rating Scale is an assessment performed by a trained rater who interviews the patient about various mood symptoms; the range=0-54, higher scores indicate more depressive symptoms, commonly accepted cut points are: 0-6 for no depression, 7-17 for mild depression, 18-24 for moderate depression, and 25 or higher for severe depression.)
  units on a scale | 19.4 (3.8) | 19.4 (3.2) | 19.4 (3.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Depressive Symptoms
Description: Change in the Hamilton Depression Rating Scale score (range=0-54, higher scores indicate more depressive symptoms), average baseline score was ~19 in both groups, and remission goal is a score of 7 or a change of ~12.
Time Frame: change from baseline at 33 weeks of gestation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Personalize Integrated Chronotherapy
Number analyzed (Participants) | 55 | 46
units on a scale | 1.6 (4.0) | 2.2 (4.5)

2. Primary Outcome: Change in Depressive Symptoms
Description: Score on the Hamilton Depression Rating Scale (range=0-54, higher scores indicate more depressive symptoms)
Time Frame: change from baseline at 36 weeks of gestation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Personalize Integrated Chronotherapy
Number analyzed (Participants) | 48 | 43
units on a scale | 3.0 (4.0) | 3.8 (5.2)

3. Primary Outcome: Change in Depressive Symptoms
Description: Score on the Hamilton Depression Rating Scale (range=0-54, higher scores indicate more depressive symptoms)
Time Frame: change from baseline at 2 weeks postpartum
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Personalize Integrated Chronotherapy
Number analyzed (Participants) | 52 | 40
units on a scale | 5.5 (5.3) | 5.8 (5.6)

4. Primary Outcome: Change in Depressive Symptoms
Description: Score on the Hamilton Depression Rating Scale (range=0-54, higher scores indicate more depressive symptoms)
Time Frame: change from baseline at 6 weeks postpartum
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Personalize Integrated Chronotherapy
Number analyzed (Participants) | 51 | 38
units on a scale | 5.2 (5.7) | 5.9 (5.4)

5. Primary Outcome: Change in Depressive Symptoms
Description: Score on the Hamilton Depression Rating Scale (range=0-54, higher scores indicate more depressive symptoms)
Time Frame: change from baseline at 18 weeks postpartum
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Personalize Integrated Chronotherapy
Number analyzed (Participants) | 47 | 37
units on a scale | 6.4 (5.0) | 7.1 (5.9)

6. Secondary Outcome: Change in Circadian Phase
Description: Time of salivary dim light melatonin onset (DLMO)
Time Frame: change from baseline at 36 weeks pregnancy
Reporting Status: Not Posted, anticipated posting 2026-04

7. Secondary Outcome: Change in Circadian Phase
Description: Time of salivary dim light melatonin onset (DLMO)
Time Frame: change from baseline at 6 weeks postpartum
Reporting Status: Not Posted, anticipated posting 2026-04

8. Secondary Outcome: Change in Sleep Timing
Description: time of sleep onset and sleep offset measured with wrist actigraphy
Time Frame: change from baseline at 33 weeks of pregnancy
Reporting Status: Not Posted, anticipated posting 2026-04

9. Secondary Outcome: Change in Sleep Timing
Description: time of sleep onset and sleep offset measured with wrist actigraphy
Time Frame: change from baseline at 36 weeks of pregnancy
Reporting Status: Not Posted, anticipated posting 2026-04

10. Secondary Outcome: Change in Sleep Timing
Description: time of sleep onset and sleep offset measured with wrist actigraphy
Time Frame: change from baseline at 2 weeks postpartum
Reporting Status: Not Posted, anticipated posting 2026-04

11. Secondary Outcome: Change in Sleep Timing
Description: time of sleep onset and sleep offset measured with wrist actigraphy
Time Frame: change from baseline at 6 weeks postpartum
Reporting Status: Not Posted, anticipated posting 2026-04

12. Secondary Outcome: Change in Sleep Timing
Description: time of sleep onset and sleep offset measured with wrist actigraphy
Time Frame: change from baseline at 18 weeks postpartum
Reporting Status: Not Posted, anticipated posting 2026-04

13. Secondary Outcome: Infant Sleep Behavior
Description: infant sleep-wake patterns will be measured with one week of ankle actigraphy
Time Frame: 18 weeks postpartum
Reporting Status: Not Posted, anticipated posting 2026-04

14. Secondary Outcome: Melatonin Levels and Timing of Onset in Breastmilk
Description: We will examine associations between salivary melatonin levels and melatonin levels in breast milk
Time Frame: 18 weeks postpartum
Reporting Status: Not Posted, anticipated posting 2026-04

ADVERSE EVENTS:
Time Frame: adverse events were assessed using the SAFTEE symptom checklist instrument at the following study visits: Visit 2 - baseline Visit 3 - 33 weeks of gestation Visit 4 - 36 weeks of gestation Visit 5 - 2 weeks postpartum Visit 6 - 6 weeks postpartum Visit 7 - 18 weeks postpartum We also collected adverse event data if participants contacted us about an AE between visits.
Arm/Group | Usual Care | Personalize Integrated Chronotherapy
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/63 | 1/57
Other Adverse Events (participants affected / at risk) | 16/63 | 16/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=63) | Personalize Integrated Chronotherapy (N=57)
hospital admission (Reproductive system and breast disorders) | 0 (0) | 1 (1) — pregnant patient was hospitalized for severe constipation requiring pain management; this was not unexpected and was deemed unrelated to the study
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=63) | Personalize Integrated Chronotherapy (N=57)
pregnancy complications (Pregnancy, puerperium and perinatal conditions) | 16 (18) | 16 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-20): https://cdn.clinicaltrials.gov/large-docs/46/NCT04364646/Prot_SAP_000.pdf